CLINICAL TRIAL: NCT04598919
Title: Use of the Src Family Kinase Inhibitor Saracatinib in the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Saracatinib in the Treatment of Idiopathic Pulmonary Fibrosis
Acronym: STOP-IPF
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Yale University (Other); Icahn School of Medicine at Mount Sinai (Other); AstraZeneca (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH); Baylor University (Other); International Center for Health Outcomes and Innovation Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5UH3TR002445 (NIH); UG3TR002445 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-10-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; Scarring of the lung; Saracatinib; randomized controlled trial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This will be a randomized (8:1 ratio), double blind, parallel design, placebo controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a randomized clinical trial, in which the patients and investigators are masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saracatinab (Active Comparator): saracatinib 125 mg once daily by mouth for 24 weeks
  Interventions: Drug: Saracatinab
- Placebo (Placebo Comparator): matching placebo once daily by mouth for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saracatinab — 125 mg once daily by mouth for 24 weeks
  Arms: Saracatinab
Drug: Placebo — once daily by mouth for 24 weeks
  Arms: Placebo

SUMMARY:
Scarring of the lung, termed pulmonary fibrosis (PF), is a chronic, progressive, and usually fatal disorder. While two anti-fibrotic drugs have been approved for treating PF of unknown cause (idiopathic pulmonary fibrosis or IPF), neither drug is curative, and nearly 40% of patients stop taking the prescribed drug within a year because of side effects. The study includes the use of saracatinib, an investigational drug originally developed to treat certain types of cancers, in the treatment of IPF in a Phase 1b/2a clinical trial.

The objectives of this study are to: i) evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics, and to explore the efficacy of saracatinib in IPF; ii) identify biomarkers of Src kinase activity and fibrogenesis linked to pulmonary fibrosis; and iii) explore the application of these biomarkers to assess the anti-fibrotic effect of saracatinib in IPF patients

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled, single-dose, four-site trial. The trial is a biomarker based, integrated Phase 1b/2a clinical trial involving 100 subjects. One group (n=50) will receive placebo, while the other group (n=50) will receive 125 mg of oral saracatinib once daily.

Randomization will be stratified by center. The randomization scheme will be in random blocks of 2 and 4 within each stratum to maintain balance. In the second part of the trial, we will use a simple randomization scheme to achieve the 8:1 randomization across sites. The study is designed to have interim analysis of the drop-out rates when approximately 30% of the randomized patients have achieved the 24-week assessment. Should the drop-out rate be higher than the 20% that is anticipated, a new sample size calculation will be performed to make sure that the power of the study is maintained at 80% .

Duration of follow-up will be 28 weeks including 24 weeks of treatment with saracatinib or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. IPF of any duration, confirmed or diagnosed by ILD center or expert according to Fleischner Guidelines (33). Subjects with a probable or indeterminant CT scan who otherwise meet the Fleischner criteria for IPF are eligible to be included in the study after a multidisciplinary evaluation. A positive Envisia genomic classifier score (34) on a lung biopsy specimen will be considered as strong evidence for a diagnosis of IPF. Subjects with a positive invisia genomic classifier score in conjunction with a probable or indeterminant CT scan are eligible to be included in the study after a multidisciplinary evaluation.
2. Women or men >40 years of age at the time of screening
3. FVC%>45% of predicted value (GLI-2012)
4. Single breath DLCO% ≥ 30 - inclusive of predicted (without bronchodilator and uncorrected for hemoglobin GLI-2017)
5. FEV1/FVC>70 (GLI-2012)
6. Provision of signed/dated written informed consent prior to any study-specific procedures
7. Females must be of nonchildbearing potential (defined as surgically sterilized [i.e., bilateral tubal ligation, bilateral oophorectomy or complete hysterectomy] or postmenopausal [defined as 12 months with no menses without an alternative medical cause] with a follicle-stimulating hormone [FSH] > 25.8 IU/L) or use a highly effective method of contraception (defined as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; progestogen only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of drug/matching placebo
8. Male subjects must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of drug/matching placebo to prevent pregnancy in a partner. Male subjects must not donate or bank sperm for the duration of the study (from the time they sign consent) and for 3 months after the last dose of drug/matching placebo.

Exclusion Criteria:

1. Requirement for supplemental oxygen > 4 L/min at rest to maintain saturation > 90%
2. Active infection at screening or randomization
3. Known active or latent hepatitis B or C
4. Life expectancy for disease other than IPF < 2.5 years (Investigator assessment)
5. Listed for lung transplantation
6. Taking pirfenidone or nintedanib in the last 4 weeks
7. Pregnancy or lactation
8. Known allergic reactions to components of saracatinib
9. Treatment with another investigational drug or other intervention within 8 weeks
10. Current smoker or tobacco use within 4 months
11. Major surgery within the past 2 months
12. Advanced hematologic, renal, hepatic, any lung disease determined by the investigator to be non-IPF related or metabolic disease that, in the opinion of the investigator, would make it unsafe for the person to receive study drug.
13. Previous lung transplantation
14. Inability to attend scheduled study visits
15. Inability to give informed consent
16. Inability to perform pulmonary function testing
17. History of malignancy in the past two years, other than squamous or basal cell skin cancer
18. Previous acute exacerbation of IPF requiring hospitalization and/or antibiotics within 90 days before the first dose of the investigational product
19. Liver function test results ≥3× upper limit of normal (ULN) liver isoform of aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT), or alkaline phosphatase (ALP) or ≥2×ULN total bilirubin (excepting documentation of benign hereditary cause). An isolated total bilirubin elevation (ie, no significant concomitant elevation in ALT or AST) at baseline of ≤ 2xULN is permitted. If there is concomitant elevation in ALT or AST to ≤3xULN, then the threshold for total bilirubin is ≤1.5xULN.
20. Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula
21. Known pulmonary hypertension (PH) requiring PH-specific treatment
22. Chronic oral corticosteroids at doses greater than prednisone 10 mg/day (or equivalent)
23. Refer to 6.5 Concomitant Therapy for exclusions based on co-medications

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of saracatinib in IPF as measured by frequency of adverse events | 24 weeks
  Safety data will be listed and summarized with patient counts and percentages in each treatment arm
Tolerability of saracatinib in IPF as measured by Severity of adverse events | 24 weeks
  A listing of all adverse events by patient will be presented. This listing will include patient number, adverse event (actual term and preferred term), event stand and end dates, CTCAE grade, relationship to the study drug/procedure, seriousness and outcome. A listing of SAEs will be produced using the similar format. This is not a scale. It is a data capture tool.
Pharmacokinetics of saracatinib in IPF as measured by serum levels | 24 weeks
  Serum levels of saracatinib
Pharmacodynamics of saracatinib in IPF as measured by change in serum β-CTX | 24 weeks
  Change in serum β-CTX as a Src kinase dependent biomarker
Efficacy of saracatinib in IPF as measured by change in FVC | 24 weeks
  Change in FVC from baseline

SECONDARY OUTCOMES:
Efficacy of saracatinib in IPF (HRCT) | 24 weeks
  Change in HRCT quantitative analysis of the extent of pulmonary fibrosis. The analysis of HRCT data will involve data-driven texture analysis (DTA), a machine learning method capable of automatic detection and quantification of lung fibrosis on HRCT
Efficacy of saracatinib in IPF (DLCO) as measured by change in DLCO | 24 weeks
  Change in diffusing capacity of the lung for carbon monoxide (DLCO)
Efficacy of saracatinib in IPF (exacerbations) as measured in time to first acute exacerbation | 24 weeks
  Time to the first acute exacerbation
Efficacy of saracatinib in quality of life in IPF (SGRQ) as measured by total score on SGRQ questionnaire | 24 weeks
  Total score on the SGRQ questionnaire. St. George's Respiratory Questionnaire (SGRQ) is a 50-item, self-administered, respiratory-specific questionnaire with items covering three domains: symptoms, activities, impacts. Each domain and a total score range from 0-100, with higher scores connoting greater impairment.
Efficacy of saracatinib in quality of life in IPF (L-IPF) as measured by total score on L-IPF questionnaire | 24 weeks
  Total score on the L-IPF questionnaire. Living with IPF (L-IPF) is an IPF-specific questionnaire whose 43 items cover two modules: symptoms and impacts. A model-based scoring algorithm has been developed via psychometric methods.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Downey, MD, Principal Investigator — National Jewish Health; Maria Padilla, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Danielle Antin-Ozerkis, MD, Principal Investigator — Yale University; Susan Mathai, MD, Principal Investigator — Baylor University Medical Center (BUMC); Annetine Gelijns, PhD, Principal Investigator — Data and Clinical Coordinating Center- InCHOIR
Locations (4):
- United States (4):
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor University Medical Center (BUMC), Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data for any analysis purpose. After the study is completed, the de-identified, archived data will be transmitted to and stored at a publicly available data repository, for use by other researchers including those outside of the study.